CLINICAL TRIAL: NCT01362088
Title: Evaluation of Sublingual Microcirculation by Means of SDF Imaging by Stepwise Ultrafiltration in CVVH Patients on the ICU
Brief Title: Microcirculation in Continuous Venovenous Hemofiltration Patients on the Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Frisius Medisch Centrum (Other)
Responsible Party: Principal Investigator, E.C. Boerma, Dr, Frisius Medisch Centrum
Other Study IDs: TPO 767
Record Dates: First submitted 2011-05-11; First posted 2011-05-27 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Continuous Venovenous Hemofiltration
Keywords: microcirculation; intensive care; ultrafiltration; CVVH

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CVVH patients

SUMMARY:
In patients where fluid is withdrawn from the bloodstream by Continuous Venovenous Hemofiltration (CVVH), the ultrafiltration rate will be calculated for a zero balance. From there, the ultrafiltration steps are performed, after increasing the ultrafiltration rate, the sublingual microcirculation is assessed by sidestream dark field (SDF). The images are subsequently randomly analyzed, and the sublingual microcirculation is expressed as a number, the microvascular flow index (MFI).

DETAILED DESCRIPTION:
Before deciding to threat a patient actively with CVVH, a target balance will be agreed for the next 12 hours. Then the ultrafiltration rate for the zero balance is calculated. From there, the ultrafiltration rate progressively increased to 50 ml per hour, up to a maximum ultrafiltration rate of 300 ml per hour.

After each increase of the ultrafiltration rate, the sublingual microcirculation is assessed by SDF.

After obtaining the desired ultrafiltration rate, the microcirculation will again be assessed before and after the patient is temporarily placed in Trendelenburg position. This could possibly show that underfill has the greatest influence on the microcirculation, and not other factors like a rising hematocrit.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 jaar
* informed consent

Exclusion Criteria:

* age < 18 jaar
* oral surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive Care patients treated with CVVH
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2011-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Difference in MFI between zero balance and maximal ultrafiltrationrate (300 ml/hr) | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Christiaan Boerma, MD, Principal Investigator — Frisius Medisch Centrum
Locations (1):
- Medical Centre Leeuwarden, Leeuwarden, Netherlands

REFERENCES:
- [Background] Bemelmans RH, Boerma EC, Barendregt J, Ince C, Rommes JH, Spronk PE. Changes in the volume status of haemodialysis patients are reflected in sublingual microvascular perfusion. Nephrol Dial Transplant. 2009 Nov;24(11):3487-92. doi: 10.1093/ndt/gfp267. Epub 2009 Jun 10. PMID 19515801